CLINICAL TRIAL: NCT06043596
Title: Evaluation of the SafeSpace App Intervention
Acronym: SafeSpace
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Child Trends (Other)
Collaborators: Power to Decide (Other); Healthy Teen Network (Other); MyHealthEd, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1309
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Health Behavior; Health Care Utilization; Unprotected Sex; Sexually Transmitted Infections
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care; Unsafe Sex; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: This research project will use an individual randomized controlled trial design in which youth recruited from social media ads will be randomized 1:1 into the experimental condition (about sexual health) and the control condition (about general health).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SafeSpace Sexual Health (Experimental): The proposed intervention is a 10-week app-based program, SafeSpace Sexual Health. SafeSpace Sexual Health will be implemented using a secure, anonymous mobile app that uses authentic stories to engage young people with sexual health information and resources. The program addresses healthy relationships, anatomy and physiology, identity, adolescent development, STIs/HIV, pregnancy and reproduction, decision-making, personal safety, communication, and accessing healthcare. Each lesson includes a story written by youth with lived experience, two to three key facts developed by sexual health experts, a reflection prompt, and two to three reputable resources.
  Interventions: Behavioral: SafeSpace Sexual Health
- SafeSpace General Health (Active Comparator): Participants in the control condition will participate in a 10-week app-based general health program, SafeSpace General Health. Lessons address general health topics including self-care, stress, sleep, nutrition, physical activity, substance use, driving and seatbelt use, and social media. Each lesson contains 2-3 key facts created by public health experts and reputable resources. Similar to SafeSpace Sexual Health, youth will receive SafeSpace General Health over 10 weeks, although SafeSpace General Health includes one lesson per week and does not contain youth stories or reflection prompts.
  Interventions: Behavioral: SafeSpace General Health

INTERVENTIONS:
Behavioral: SafeSpace Sexual Health — The overall goal of the program is to prevent adolescent pregnancy and STIs by increasing sexual agency, increasing the use of condoms and contraception, and promoting healthy relationships and healthy life skills among adolescents.
  Arms: SafeSpace Sexual Health
Behavioral: SafeSpace General Health — This arm represents the comparison group. SafeSpace General Health will act as the active comparator, while providing youth with lessons, facts, and resources about general health topics.
  Arms: SafeSpace General Health

SUMMARY:
The goal of this study is to evaluate the impact of SafeSpace Sexual Health App, an innovative sexual health promotion program focused on reducing sexual risk factors and promoting sexual and reproductive health and wellbeing among young people assigned female or intersex at birth, particularly Black and/or Latine youth, LGBTQ+ youth, youth in states with high teen birth rates and youth who live in rural communities. This study utilizes a two-arm randomized control trial design to measure impacts of receiving the SafeSpace Sexual Health program compared to receiving a similar-length control app program, SafeSpace General Health that focuses on general health.

The investigators will ask participants to:

* Keep the SafeSpace app downloaded to their device and visit the app regularly over the course of 10 weeks.
* Provide contact information.
* Receive and open app push notifications for 10 weeks (up to 3 per week).
* Complete 3 online surveys over a year: baseline, short-term follow-up (10 weeks after baseline), and long-term follow up (9 months after short-term follow-up).
* Receive occasional text messages from the study team.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be assigned female or intersex at birth
* Participants must be youth in the U.S. (14-18 years old)
* Participants must have daily access to an iPhone

Exclusion Criteria:

- Participants must not be currently pregnant or currently trying to become pregnant

Other Criteria:

- The study's priority/preference population is for Black and/or Latine youth, LGBTQ+ youth, youth from geographic areas with high teen birth rates, and youth living in rural areas.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Penile-vaginal sex without a condom or a more effective method of contraception | Past 3 months at baseline; past 9 months at long-term follow-up
  Yes = Had penile-vaginal sex without using pill, shot, patch, ring, IUD, implant, or condom every time; No = Did not have penile-vaginal sex OR always used pill, shot, patch, ring, IUD, implant, or condom during penile-vaginal sex

SECONDARY OUTCOMES:
Penile-vaginal sex or anal sex without a condom every time | Past 3 months at baseline; past 9 months at long-term follow-up
  Yes = Had penile-vaginal sex or anal sex without using a condom every time OR had anal sex without use of a condom every time.
  No = No penile-vaginal sex AND no anal sex; or No = No penile-vaginal sex AND condom use during anal sex every time; or No = condom use during every penile vaginal sex AND no anal sex
Utilization of sexual health services | Has received SRH services in the past 12 months or has an appointment scheduled in the next 3 months at baseline; Received SRH services in the past 9 months or has an appointment scheduled in the next 3 months at long-term follow-up.
  Yes = has seen a health care provider (clinic or doctor's office) for any sexual or reproductive health services in the past 12 months No = did not see a health care provider for SRH services in the past 12 months
Number of Sexual and Reproductive Health topics discussed with a trusted adult in the past 3 months. | Past 3 months at baseline; past 10 weeks at short-term follow-up; past 9 months at long-term follow-up
  Score of talking with trusted person in the past 3 months about topic categories including either sexual orientation or gender identity; when to have sex; receiving SRH services; STIs and contraception; consent or pleasure in the past 3 months. For this scale, there is a minimum score of 0 and a maximum score of 7 with a higher score indicating a better outcome
Sexual agency during every recent sexual experience or no recent sexual experiences | Past 3 months at baseline; past 10 weeks at short-term follow-up; past 9 months at long-term follow-up
  Dependent on the frequency of a) communicating with their partners(s) about what they like, dislike, or want to try, b) asking their partner(s) what they like, dislike, or want to try, and c) asking or giving consent to their partner(s). Those who haven't engaged in sexual activity within the relevant time frame will be considered to have sexual agency

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Manlove, PhD, Study Director — Child Trends; Elizabeth L Cook, MSPH, Study Director — Child Trends; Riley Steiner, PhD, Principal Investigator — Power to Decide
Locations (1):
- Child Trends, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No